CLINICAL TRIAL: NCT03940690
Title: Multicenter Randomized Controlled Trial on the Interest of Intravitreal Injections of Anti-VEGF as Initial and Adjuvant Treatment in Coats Disease
Brief Title: Interest of Intravitreal Injections of Anti-VEGF as Initial and Adjuvant Treatment in Coats Disease
Acronym: COATS-VEGF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study futility based on the interim analysis
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FME_2018_9
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Retinal Telangiectasis; Coats Disease
Keywords: Retinal Telangiectasis; Coats Disease; Anti-VEGF (Vascular Endothelial Growth Factor)
MeSH Terms: conditions — Retinal Telangiectasis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-VEGF injections (bevacizumab) (Experimental): 5 anti-VEGF injections of bevacizumab at months 0, 1, 2, 4 and 6, combined with laser at months 2, 4 and 6 (laser optional at month 9
  Interventions: Drug: Anti-VEGF injections of bevacizumab
- Arm : laser only (Active Comparator): 3 sessions of laser at months 0, 1 and 2, completed if needed with laser at months 4, 6 et and 9
  Interventions: Device: Laser

INTERVENTIONS:
Drug: Anti-VEGF injections of bevacizumab — 5 anti-VEGF injections of bevacizumab at months 0, 1, 2, 4 and 6, combined with laser at months 2, 4 and 6 (laser optional at month 9)
  Arms: Anti-VEGF injections (bevacizumab)
Device: Laser — 3 sessions of laser at months 0, 1 and 2, completed if needed with laser at months 4, 6 et and 9
  Arms: Arm : laser only

SUMMARY:
Coats disease is a predominantly unilateral progressive retinal vascular disease, characterized by retinal telangiectasias with intra- or subretinal exudate deposits, which can lead to retinal detachment and one-sided blindness. Several treatment modalities are available and the choice of one of them depends on the stage of the disease and the habits of each center (laser photocoagulation, cryotherapy ...). VEGF (Vascular Endothelial Growth Factor) was found to be significantly elevated in the aqueous humor and subretinal fluid of patients with Coats disease. Several studies have shown the potential efficacy of intra-vitreous injections of anti-VEGF. But the results on their effectiveness have been evaluated only on small series of patients. Most published studies have analyzed their efficacy combined with another treatment, mainly laser photocoagulation. The true efficacy of anti-VEGF therapy as initial therapy, and then combined in Coats disease remains unknown. Currently, several centers are initiating first-line anti-VEGF injections, although no rigorous evaluation of this therapeutic strategy has been conducted.

The identification of the best treatment regimen will allow in the future the reduction of laser reprocessing and will ensure a better functional benefit in the affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Coats disease confirmed by fundus examination and fluorescein angiography
* Stage 2 or 3 at the fundus (Shields classification)
* Naive to any eye treatment on the eye affected by Coats disease

Exclusion Criteria:

* Other ocular pathology on the eye affected by Coats' disease
* Bilateral forms of the disease
* History of hypersensitivity to bevacizumab
* History of hypersensitivity to products of Chinese hamster ovary cells or other recombinant human or humanized antibodies
* Allergic reaction in a previous fluorescein retinal angiogram
* Pregnancy or breastfeeding
* Active or suspected periocular infection
* Contraindication to treatments used for general anesthesia and morphine derivatives
* Cardiovascular, haemorrhagic and gastrointestinal risks
* Premature baby who has not reached the correct age of 37 weeks

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with improvement of stage of disease, according to the Shields classification | 6 months after randomization
  Stages assessed by retinal multimodal imaging (retinophotography, optical coherence tomography when age allows, retinal fluorescein angiography) by two independent expert ophthalmologists

CONTACTS AND LOCATIONS:
Overall Officials: Florence METGE, Principal Investigator — fmetge@for.paris
Locations (6):
- France (6):
  - Centre hospitalier René Dubos (Pontoise), Cergy-Pontoise, France
  - Hôpital Universitaire Necker Enfants Malades, APHP, Paris, France
  - Fondation Ophtalmologique A. de Rothschild, Paris, France
  - CHU de Reims, Reims, France
  - Clinique Rive Gauche, Toulouse, France
  - CHU de Bordeaux, Bourdeaux

IPD SHARING:
Plan to Share IPD: Undecided